CLINICAL TRIAL: NCT00705354
Title: Pilot Study To Evaluate A Pharmacologically Active Nasal Sponge Following
Brief Title: Pilot Study To Evaluate A Pharmacologically Active Nasal Sponge Following Endoscopic Sinus Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left the institution requested termination.
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-119
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Sinusitis; Chronic Sinusitis
Keywords: Sinusitis; Chronic Sinusitis; Nasal Surgery; Functional Endoscopic Sinus Surgery (FESS); Enoscopic Sinus Surgery (ESS)
MeSH Terms: conditions — Sinusitis | interventions — Bacitracin; Anti-Bacterial Agents; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Control group undergoing standard ESS will have a saline soaked Nasopore sponge placed during surgery and will receive routine oral antibiotics post-operatively
  Interventions: Procedure: Nasopore sponge soaked with saline
- 2 (Experimental): Treatment group undergoing ESS will have Nasopore sponge soaked with Bacitracin, but will not receive oral antibiotics post-operatively
  Interventions: Drug: Bacitracin

INTERVENTIONS:
Drug: Bacitracin — Nasopore sponge soaked with Bacitracin, placed in middle meatus of the nose. No post-op oral antibiotics
  Other Names: ESS; Endoscopic Sinus Surgery; Nasopore; Anti-Bacterial
  Arms: 2
Procedure: Nasopore sponge soaked with saline — Nasopore sponge soaked with saline placed during surgery and will receive routine oral antibiotics post-operatively
  Other Names: ESS; Endoscopic Sinus Surgery; Nasopore
  Arms: 1

SUMMARY:
This study will compare the incidence of post-op infection after sinus surgery using conventional post-op oral antibiotics to the incidence of infection after sinus surgery when a bio-resorbable antibiotic soaked nasal sponge is used in the nasal cavity in lieu of post-op oral antibiotics. The nasal sponge is a routine nasal dressing used after sinus surgery and will therefore be placed in all patients.

DETAILED DESCRIPTION:
Sinusitis affects 37 million people each year making it one of the most common health problems in the United States. It has a large impact in direct healthcare expenditures, significant loss of workplace productivity and a greater impact on quality of life than diabetes or congestive heart failure.

The most frequently used treatments are medications and/or Functional Endoscopic Sinus Surgery(FESS). 100 subjects undergoing ESS will participate, randomized into two groups, treatment and control. All subjects will have a Nasopore sponge placed into the middle meatus of the nose at the end of the procedure(The sponge is FDA approved and commonly used. Subjects in the treatment group will receive a Nasopore sponge soaked in Bacitracin solution. These subjects will not receive oral antibiotics post-operatively. The control group subjects will have a saline soaked Nasopore sponge laced during surgery and will receive routine oral antibiotics post-operatively. The hypothesis is that subjects who receive the antibiotic soaked nasal sponge in lieu of saline soaked nasal sponge will have infection rates comparable to those who receive systemic antibiotics, but because they will not receive systemic antibiotics, the treated group will have fewer side effects and the cost to treat them will be less.

ELIGIBILITY:
Inclusion Criteria:

* Subjects requiring Endoscopic Sinus Surgery

Exclusion Criteria:

* Pediatric subjects <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The two groups of subjects will be compared on clincal & demographic characteristics. Evaluation of any new infection (no or yes). | Post surgical evaluations at 2/3 weeks and 3 months

SECONDARY OUTCOMES:
Clinical and demographic data will be evaluate presence/absence of inflammation of surrounding, adhesions, pain, granulation tissue | Evaluated at 2/3 weeks and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Catalano, M.D., Principal Investigator — Lahey Clinic, Inc.
Locations (1):
- Lahey Clinic, Inc., Burlington, Massachusetts, United States

REFERENCES:
- [Background] Catalano PJ, Roffman EJ. Evaluation of middle meatal stenting after minimally invasive sinus techniques (MIST). Otolaryngol Head Neck Surg. 2003 Jun;128(6):875-81. doi: 10.1016/S0194-59980300469-8. PMID 12825040